CLINICAL TRIAL: NCT05776095
Title: A Prospective, Multicenter Study to Evaluate Safety and Performance Outcomes of Eyedeal Intraocular Lens Implantation After Cataract Removal
Brief Title: Evaluation of Safety and Performance Outcomes of Eyedeal IOL Implantation After Cataract Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Eyedeal Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-301
Record Dates: First submitted 2023-02-17; First posted 2023-03-20 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Lens Implantation, Intraocular
Keywords: Cataract; Intraocular lens; IOL
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, two-center interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyedeal® IOL (Experimental): Eyedeal® Model PX65AS1 IOL
  Interventions: Procedure: Cataract surgery; Device: Eyedeal® Model PX65AS1 IOL

INTERVENTIONS:
Procedure: Cataract surgery — Subjects will undergo surgery to remove cataract (the cloudy lenses) via phacoemulsification, and implant the Eyedeal® Model PX65AS1 IOL in the eye capsule.
Device: Eyedeal® Model PX65AS1 IOL — Subjects will undergo surgery to remove cataract (the cloudy lenses) via phacoemulsification, and implant the Eyedeal® Model PX65AS1 IOL in the eye capsule.

SUMMARY:
A cataract is the clouding of the natural lens in the eye and is very common as when getting older. A cloudy lens makes it difficult to see. A cataract is treated by removing the cloudy lens and replacing it with an intraocular lens (known as an IOL). The goal of this clinical trial is to determine if the Eyedeal® IOL can be safely implanted in a subject's eye and if it can replace efficiently the natural lens.

Subjects will be asked to attend a total of seven visits for this study for a period of 12 months after surgery.

DETAILED DESCRIPTION:
To investigate the safety and performance of the Eyedeal® PX65AS1 intraocular lens (IOL)

* To evaluate the safety profile with regards to best-corrected visual acuity, and adverse events
* To evaluate the performance with regards of best corrected distance VA after the device implantation

The Eyedeal® IOL (PX65AS1) is a foldable single-piece ultra-violet absorbing posterior chamber intraocular lens (IOL). It is an optical implant to replace the human crystalline lens in the visual correction of aphakia in adult patients after cataract removal. The Eyedeal® PX65AS1 IOL lens is made of a high refractive index soft cross-linked polyolefin. The Eyedeal® PX65AS1 IOL lens has an aspheric optic with symmetric optic design and spherical neutral and correct lens's own spherical aberration supporting haptics to provide proper position of the IOL optic within the capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (22 years of age or older at the time of surgery) of any gender and race, diagnosed with age related cataracts in one eye.
2. Preoperative best corrected distance visual acuity (BCDVA) of 20/32 or worse.
3. Projected postoperative BCDVA 0.20 logMAR or better in the study eye, as determined by Investigator's medical judgment.
4. Calculated spherical power targeted at emmetropia at distance in the study eye.
5. Calculated lens power within the available range for the Eyedeal® Model PX65AS1 IOL (+0.50D - +34.00D).
6. Planned cataract removal by phacoemulsification procedure.
7. Clear intraocular media other than cataract, in the study eye.
8. Pharmacologically dilated pupil size of at least 6.0mm.
9. 2.0 D or less of preoperative astigmatism in the study eye.
10. Willing and able to complete all required postoperative visits.
11. Able to comprehend and sign or through a representative, with a witness present, a statement of IRB or EC approved Informed Consent Form (ICF).

Exclusion Criteria:

1. Any type of cataract (e.g., traumatic, congenital, polar) other than those noted in inclusion criteria.
2. Ocular conditions which could affect the stability of the IOL (e.g., pseudoexfoliation, zonular dialysis, evident zonular weakness or dehiscence, etc.) in the study eye.
3. Any anterior segment pathology likely to increase the risk of complications from phacoemulsification cataract extraction (e.g., chronic uveitis, iritis, iridocyclitis, aniridia, rubeosis iridis, clinically significant corneal disorders, (Fuch's, or anterior basement membrane dystrophy, etc.) in the study eye.
4. Mature cataract that is likely to prolong phacoemulsification and/or lead to intraoperative complications prior to attempted IOL implantation.
5. Any visually significant intraocular media opacity other than cataract in the study eye.
6. History of any clinically significant retinal pathology or ocular diagnosis (e.g., diabetic retinopathy, ischemic disease, macular degeneration, retinal detachment, amblyopia, optic neuropathy, microphthalmos, aniridia, neuro-ophthalmic disease, fixation problems etc.) in the study eye that could alter or limit final postoperative visual prognosis.
7. History of any intraocular, retinal, corneal or refractive surgery in the study eye (including LASIK, PRK, LRI, etc.).
8. History of cystoid macular edema in the study eye.
9. History of serious corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.) in either eye.
10. Severe dry eye that, in the opinion of the investigator, would impair the ability to obtain reliable study measurements.
11. Uncontrolled glaucoma and/or optic atrophy in the study eye.
12. Subjects with large refractive errors (hyperopia/myopia) of axial or pathologic origin that, in the opinion of the investigator, could confound outcomes.
13. Abnormal corneal findings in either eye (e.g. keratoconus, pellucid marginal degeneration, or irregular astigmatism).
14. Uncontrolled systemic disease (e.g., diabetes mellitus, active cancer treatment, mental illness, etc.) in the opinion of the investigator, would put the subject's health at risk and/or prevent the subject from completing all study visits.
15. Systemic medication that, in the opinion of the investigator, may confound the outcome or increase the intraoperative and post-operative risk to the subject (e.g., tamsulosin hydrochloride) or other medications including anticholinergics, alpha adrenergic blocking agents with similar side effects (e.g., small pupil/floppy iris syndrome).
16. Subjects who may reasonably be expected to require any additional ophthalmic surgical intervention at any time during the study (other than YAG capsulotomy).
17. Need for concomitant procedures (e.g., glaucoma surgery, LRI, RK, LASIK, etc.).
18. Fellow eye BCDVA worse than 1.0 logMAR.
19. Extremely shallow anterior chamber (< 2.0 mm).
20. Participation in any other drug or device clinical trial within 30 days prior to enrolling this study and/or during study participation.
21. Pregnancy or lactation.
22. Subject who, in the judgment of the clinical investigator, is not suitable for participation in the study for any clinical reason, as documented by the investigator on the patient's Case Report Forms - CRFs).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
EFFICACY OUTCOME MEASURE - Uncorrected Distance Visual Acuity | 12 months
  Uncorrected distance Visual Acuity is measured in accordance with ISO 11979-7:2018 - Appendix E: BCVA 20/40 or better in 95% of cases. The stability and consistency of visual results will be measured over time.
SAFETY OUTCOME MEASURE - Best Corrected Visual Acuity | 12 months
  The safety of the Eyedeal® Model PX65AS1 IOLs (Xi'an Eyedeal Medical Technology Co., Ltd.) will be measured by the following criteria:
  Loss of BCDVA measured in accordance with ISO 11979-7:2018-Appendix E
SAFETY OUTCOME MEASURE - Evaluation of Patient record | 12 months
  The safety of the Eyedeal® Model PX65AS1 IOLs (Xi'an Eyedeal Medical Technology Co., Ltd.) will be measured by the following criteria:
  Patient record of inflammation, discomfort, or pain following surgery related to the Eyedeal® Model PX65AS1 IOL (Xi'an Eyedeal Medical Technology Co., Ltd.) .
  .
SAFETY OUTCOME MEASURE - Evaluation of Adverse Events | 12 months
  The safety of the Eyedeal® Model PX65AS1 IOLs (Xi'an Eyedeal Medical Technology Co., Ltd.) will be measured by the following criteria:
  Evaluation of all adverse events, adverse device effects and device deficiencies at post-operative examinations

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Auffarth, Prof, Principal Investigator — University Eye Clinic Heidelberg
Locations (2):
- University Eye Clinic Heidelberg, Heidelberg, Baden-Wurttemberg, Germany
- Department of Ophthalmology, Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Lithuania